CLINICAL TRIAL: NCT01846286
Title: Molecular Epidemiology of Neuropathic Pain in Head and Neck Cancer
Brief Title: Neuropathic Pain in Head and Neck Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2012-0642; 1R01DE022891 (NIH)
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Head and Neck Cancer
Keywords: Neuropathic Pain; Squamous cell cancer of the head and neck; acute pain; pain management; genome-wide analyses; Squamous cell carcinoma of the head and neck; chronic pain; neuropathic; locoregional squamous cell carcinoma of the head and neck
MeSH Terms: conditions — Head and Neck Neoplasms; Neuralgia; Acute Pain; Agnosia; Squamous Cell Carcinoma of Head and Neck; Chronic Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newly Diagnosed HNC: For AIM 2 and AIM3, Newly diagnosed and previously untreated patients with locoregional squamous cell carcinoma of the head and neck recruited at MD Anderson: Pain assessed at baseline, weekly during treatment, and during clinic visits (every 6-8 weeks) for a period of 3 months after treatment. Quantitative sensory testing performed at baseline and at 3 months from completion of treatment to determine nociceptive versus neuropathic component.
  Interventions: Behavioral: Questionnaires; Other: Quantitative Sensory Testing

INTERVENTIONS:
Behavioral: Questionnaires — Five questionnaires about pain and symptoms, each taking approximately 25 - 50 minutes to complete
  Other Names: Surveys
Other: Quantitative Sensory Testing — Tests measure sensitivity to touch, coolness, warmth, hot/cold feeling, and pin pricks. The sensory tests will take about 30 minutes to 1 hour to complete.
  Other Names: QST

SUMMARY:
The goal of this research study is to learn more about chronic pain associated with cancer treatment.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will complete the following tests and procedures at the beginning and at the end of the study (on clinic visits, typically around 3-6 months after completion of treatment):

°You will complete 5 questionnaires about any pain and other symptoms you may have had, your general well-being, drugs you may be taking, and personal information, such as your age. The questionnaires will take about 25-50 minutes to complete.

Every week during treatment period, you will complete a questionnaire about pain you may be having. This questionnaire will take about 5-10 minutes to complete.

Length of Study:

You will be on study for about 3-6 months after the last day of treatment.

This is an investigational study. Up to 1200 will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Aim 1 Discovery Phase: The samples are from a large NIH-funded Genome-wide association study of squamous cell carcinoma of the head and neck (Shete; PI). A total of 2900 "case" patients and 1200 control patients were recruited for the study. In this study, we will only use cases who were: a) Newly diagnosed, untreated, histopathologically confirmed squamous cell carcinoma of the oral cavity, pharynx, or larynx; b) No previous cancers; c) Age 18 years or older; d) white Caucasian.
2. Aim 2: a) Newly diagnosed patients (have not had any prior cancer treatment) with loco-regional squamous cell carcinoma of the head and neck, b) Will receive cancer treatment at MDACC or at Ben Taub, c) Are 18 years or older, d) English or Spanish speaking; e) Able to understand the description of the study and give written informed consent; f) Will state that they will receive follow-up at MD Anderson post-treatment or at Ben Taub. This sample will also be included in the Validation Phase of Aim 1. We note that population stratification, i.e., the presence of a systematic difference in allele frequencies between subpopulations in a population possibly due to different ancestry, is an issue for genetic association studies.
3. Aim 3: Patients included in aims 1 and 2.

Exclusion Criteria:

1) Exclusion for Aim 2: a) Patients with distant metastasis (Stage IVC); b. Patients participating in clinical trials/ investigational drugs for pain control. Aim 1 (discovery phase) and Aim 3 will use existing data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For AIM 1: Squamous cell carcinoma of the head and neck patients for whom genome-wide (730,525 SNPs) and pain data are available; AIM 2: Newly diagnosed and previously untreated patients with locoregional (excludes Stage IVc) squamous cell carcinoma of the head and neck recruited at the Head and Neck Center at MD Anderson; AIM 3: Populations from AIM 1 & 2.
Sampling Method: Non-Probability Sample
Enrollment: 838 (Actual)
Dates: Start 2012-10-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Genome-wide analyses on Participants with squamous cell carcinoma of the head and neck | 5 years
  Genome-wide analyses, 730,525 Single Nucleotide Polymorphisms (SNPs), on participants with squamous cell carcinoma of the head and neck in order to identify potentially novel gene variants associated with the development of chronic pain (neuropathic versus nociceptive).

SECONDARY OUTCOMES:
Assessed Pain Severity (mean pain) | Baseline to 3 months post treatment
  Pain Severity determined using 0-10 numeric rating scale (0= 'no pain' and 10='worst pain imaginable'). Pain assessed at baseline (start of the study), weekly during treatment, and during clinic visits (every 6-8 weeks) for a period of 3 months after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Cielito C. Reyes-Gibby, MSN, DRPH, Study Chair — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Lyndon B. Johnson General Hospital (LBJ), Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org